CLINICAL TRIAL: NCT00369109
Title: Collection of Skin Biopsy With Hair Follicles as Surrogate to Develop Biomarker Assays From Patients With Advanced Solid Tumor Malignancies Receiving Either Single Agent Weekly Irinotecan or Gemcitabine
Brief Title: Skin Biopsies and DNA Analysis in Patients Receiving Irinotecan or Gemcitabine For Advanced Solid Tumors
Status: Completed | Type: Observational
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000479118; P30CA022453 (NIH); WSU-2005-039; ZENECA-D1040M00003; WSU-0512003224
Record Dates: First submitted 2006-08-24; First posted 2006-08-29 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Breast Cancer; Colorectal Cancer; Pancreatic Cancer
Keywords: recurrent colon cancer; stage III colon cancer; stage IV colon cancer; recurrent rectal cancer; stage III rectal cancer; stage IV rectal cancer; recurrent pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer; stage IV pancreatic cancer; recurrent breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Pancreatic Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Immunohistochemistry; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: biologic sample preservation procedure
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Procedure: biopsy

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors identify and learn more about biomarkers related to cancer.

PURPOSE: This laboratory study is collecting skin biopsy specimens from patients receiving irinotecan or gemcitabine for advanced solid tumors and using them to study change in DNA due to this treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the level of p-Chk1 and phospho-histone 2AX (p-H2AX), an indicator of DNA damage, and possibly downstream pathway markers in hair follicles from skin biopsies of patients treated with gemcitabine hydrochloride or irinotecan hydrochloride for advanced solid tumors.

Secondary

* Characterize the method for measurement (immunohistochemistry).
* Measure inter- and intra-patient variability for the biomarker.
* Partially characterize the dynamic time course of p-Chk1 and p-H2AX after administration of a DNA-damaging agent.

OUTLINE: This is a multicenter study.

Patients undergo collection of 2 skin biopsies with hair follicles at 4 and 8 hours or at 4 and 6 hours after the start of irinotecan hydrochloride or gemcitabine hydrochloride treatment on day 1 of course 1. Repeat biopsies will be taken at 4, 6, or 8 hours after the start of irinotecan hydrochloride or gemcitabine hydrochloride on day 1 of 2 successive courses.

Tissue is examined by immunohistochemistry and possibly other methods for changes in p-Chk1 and pH2AX.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of advanced solid tumor malignancy (preferably colorectal, pancreatic, or breast cancer)
* Scheduled to receive a standard dose, weekly regimen of either irinotecan hydrochloride or gemcitabine hydrochloride

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* No DNA-damaging agent within the past 13 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-02; Primary Completion 2006-11 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Level of p-Chk1 and phospho-histone 2AX (p-H2AX) and possibly downstream pathway markers in hair follicles from skin biopsies of patients treated with gemcitabine hydrochloride or irinotecan hydrochloride for advanced solid tumors

SECONDARY OUTCOMES:
Characterization of the method for measurement (immunohistochemistry)
Inter- and intra-patient variability for the biomarker
Dynamic time course of p-Chk1 and p-H2AX after administration of a DNA-damaging agent

CONTACTS AND LOCATIONS:
Overall Officials: Patricia M. LoRusso, DO, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (2):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States
- Christie Hospital NHS Trust, Manchester, England, United Kingdom